CLINICAL TRIAL: NCT06424327
Title: Pulmonary Segmentectomy for Lung Cancer: A Real-World International Registry-TSOG 108
Brief Title: A Registry for People With Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 24-127
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Lung Cancer Stage I
Keywords: lung cancer; lung cancer stage 1; segmentectomy; Memorial Sloan Kettering Cancer Center; 24-127
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Lung Cancer: Participants undergoing planned pulmonary segmentectomy for primary lung cancer
  Interventions: Other: Patient-Reported Outcomes Measurement Information System

INTERVENTIONS:
Other: Patient-Reported Outcomes Measurement Information System — Participants-reported outcomes will be collected using the Patient-Reported Outcomes Measurement Information System (PROMIS). PROMIS is a web-based platform developed by the National Institutes of Health. Scoring is standardized on a scale from 0 to 100, with a population mean of 50 and standard deviation of 10 units. High scores mean more of the concept being measured. This study will use PROMIS surveys assessing three domains: physical function (PROMIS bank version 2.0), pain interference (PROMIS bank version 1.1), and dyspnea severity (PROMIS bank version 1.0)
  Other Names: PROMIS

SUMMARY:
Participants will complete questionnaires before surgery, between 2 to 4 weeks after surgery, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical Stage I with suspected NSCLC, classified preoperatively based on the AJCC TNM staging manual, 9th edition o Note: Tissue diagnosis of NSCLC is not required before enrollment. A pathologic diagnosis of NSCLC may be confirmed preoperatively with biopsy, intraoperatively with frozen section, or postoperatively on final pathology

Exclusion Criteria:

* Actively receiving lung cancer treatment or a history of lung cancer in the previous 5 years
* History of chemotherapy or radiation therapy for a previous lung cancer
* Synchronous secondary cancer in the lung or elsewhere in the body at the time of surgery
* Carcinoid tumors
* History of other malignancies within the past 3 years, with the exception of non-melanoma skin cancer, superficial bladder cancer, and carcinoma in situ of the cervix
* Actively receiving treatment for other malignancies
* Cases of lobectomy in conjunction with segmentectomy from another lobe and ≥2 segmentectomies from different lobes either en bloc or separate will be excluded from the primary analysis.

  * Multi-segmental resection from the same lobe is not a criterion for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study subjects will be recruited from their respective clinics (i.e., Thoracic Surgery, Pulmonary, Survivorship, etc.) at participating sites. Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team by screening patients' medical records. If eligible, the study will be discussed with each patient.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2029-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Determine 3-year disease-free survival/DFS among patients undergoing pulmonary segmentectomy for lung cancer. | 3 years
  DFS is measured from the date of surgery to the date of recurrence or death
Determine 5-year disease-free survival/DFS among patients undergoing pulmonary segmentectomy for lung cancer. | 5 years
  DFS is measured from the date of surgery to the date of recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: David Jones, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (14):
- United States (12):
  - Rush University Medical Center (Data collection only), Chicago, Illinois
  - Endeavor Health, Evanston, Illinois
  - University of Michigan (Data Collection Only), Ann Arbor, Michigan
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - ALLEGHENY HEALTH NETWORK (Data Collection Only), Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center (Data Collection Only), Houston, Texas
- Canada (2):
  - University Health Network (Data Collection Only), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montreal (Data Collection Only), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org